CLINICAL TRIAL: NCT07380815
Title: Assessment of Physical Activity During Radiation Therapy for LUNG Cancer
Brief Title: Physical Activity During Radiation Therapy for Lung Cancer
Acronym: APART-LUNG
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Other Study IDs: APART-LUNG
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prospective Study
Keywords: lung cancer; radiation therapy; physical activity
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with steps counted by their smart phone: The purpose is to obtain a patient's mean number of steps per week during week 1 and week 5 of a radiation therapy course for lung cancer directly from the patient's smart phone which has a step counter.

SUMMARY:
The primary objective of this trial is to evaluate patterns of physical activity during radiation therapy for lung cancer and to estimate the within-patient change in physical activity between Week 1 and Week 5 of radiation therapy, measured by smart phone-recorded step counts normalized for device carrying time. The trial is exploratory in nature with the aim to generate scientific hypotheses to be investigated in future clinical trials.

DETAILED DESCRIPTION:
Lung cancer belongs to the most common types of solid cancer in Europe and Northern America. A considerable number of patients with lung cancer receive conventionally fractionated radiation therapy with or without systemic treatment. Radiation therapy may be associated with adverse events affecting healthy tissues within the radiation field but also with fatigue and a decreased level of physical activity or function. Patients who experience significant treatment-related toxicity may not be able to receive the complete radiation therapy as planned. Maintaining or even improving the level of activity by physical exercise or walking a certain number of steps per day may be helpful in this context. A benefit of exercise has been suggested in a retrospective study of 184 cancer patients receiving neoadjuvant chemotherapy, including 31 patients with lung cancer. Adherence to an exercise program was associated with fewer dose reductions and delays of chemotherapy. Moreover, several studies performed in patients with lung cancer suggested that physical activity had a positive effect on the patient's quality of live. Thus, physical activity prior to and during chemo- and/or immunotherapy for lung cancer appears important. This may also be true for patients with lung cancer treated with radiation therapy. However, adherence to an exercise program sometimes may be challenging for the patients, particularly if they experience treatment-related fatigue or other adverse events. The question arose whether an easy-to-use mobile app installed on the patient's smart phone reminding patients several times daily to perform a certain number of steps will have a positive effect on their physical activity during a course of radiation therapy. Such an app is planned to be tested in a prospective trial. However, step counts derived from smart phones are influenced by variability in device carrying time, as patients may not carry their phones consistently throughout the day. This variability introduces measurement heterogeneity that must be explicitly addressed in the statistical design and analysis. The present study is designed as a pilot investigation for this prospective trial to evaluate changes in physical activity during radiation therapy while establishing a robust and Good Clinical Practice (GCP)-compliant analytical framework for smart phone-derived step data. Physical activity is assessed during Week 1 and Week 5 of radiation therapy using a smart phone application. A total of approximately 20 patients qualifying for the Full Analysis Set are planned to be enrolled and documented. Recruitment of all patients should be completed within 3 months. This period also represents the total running time for this study. The study is designed as a pilot and feasibility investigation and is not intended to provide confirmatory evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven lung cancer
2. Treatment with ≥50 Gy of conventionally fractionated radiation therapy
3. Possession of and ability to use a smart phone plus a step counter
4. Age ≥18 years
5. Written informed consent
6. Capacity of the patient to consent

Exclusion Criteria:

1. Expected Non-Compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received conventionally fractionated radiation therapy for lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean number of steps per week during week 1 and week 5 of radiation therapy for lung cancer | through study completion, 5 weeks
  The primary endpoint is to assess the within-patient difference in weekly average steps per wear-hour of the smart phone (Week 5 minus Week 1 of radiation therapy). Any type of smart phone is allowed, as long as it has a step counter.

SECONDARY OUTCOMES:
Wear-time of the smart phone | through study completion, 5 weeks
  The mean wear-time of the smart phone per day (given in hours) during week 1 and week 5 of the radiation therapy course is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, Principal Investigator — University of Luebeck

IPD SHARING:
Plan to Share IPD: No